CLINICAL TRIAL: NCT03808480
Title: Nivolumab After Cyclophosphamide and Doxorubicin(CA) Induction Therapy in Previously Treated Advanced Non-squamous Cell Non-small Cell Lung Cancer With PD-L1<10%
Brief Title: Nivolumab After Cyclophosphamide and Doxorubicin Induction Therapy in NSCLC With PD-L1<10%
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji-youn Han, Principle Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2018-0267
Record Dates: First submitted 2018-12-26; First posted 2019-01-17 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CA and Nivolumab (Experimental): After 1 cycle of cyclophosphamide and doxorubicin (CA) induction therapy, Nivolumab 360mg flat dose will be given on day 1 with CA chemotherapy in a 21-day cycle.
  After the completion of 4 cycles of CA chemotherapy, Nivolumab will be continued as a single agent at a dose of 480mg flat dose every 4 weeks until loss of clinical benefit
  Interventions: Drug: CA and Nivolumab

INTERVENTIONS:
Drug: CA and Nivolumab — Cyclophosphamide 500mg/m2 IV on D1 (C1-4), 1cycle=21days) Doxorubicin 50mg/m2 IV on D1 (C1~4, 1cycle=21days) Nivolumab 360 mg/IV C2~4 D1 (1cycle=21days) Nivolumab 400mg/IV on D1 from Cycle 5 every 4 weeks.
  Other Names: Opdivo

SUMMARY:
Nivolumab is now the standard of care for second-line treatment of advanced squamous or nonsquamous NSCLC regardless of the tumor's expression of PD-1L. CheckMate057 trial results showed that in unselected patients with advanced or recurrent nonsquamous NSCLC who had stopped responding to a platinum-based chemotherapy regimen, treatment with nivolumab produced significantly better overall survival during follow-up as long as 18 months, compared with a docetaxel-based regimen. But during the first 3 months on randomized treatment, 15 more patients died in the nivolumab arm than in the docetaxel arm. This quickly reversed during months 4-6 on treatment, when nine more patients died on docetaxel than on nivolumab. A post hoc analysis showed a trend to a higher risk for death during the first 3 months of nivolumab treatment among patients with poorer prognostic features, more aggressive disease, and low or no tumor expression of PD-L1. In addition, only a subgroup of patients benefits from nivolumab with response rates of 20% in unselected cohorts and 10% in low PD-L1 expression cohort. Strategies to render the tumor micro-environment (TME) more susceptible to anti-PD1 might include stimulation of anti-cancer immune responses by induction treatment with low dose chemotherapy.

Given the potent immune-modulating effects and anti-tumor activity of cyclophosphamide and doxorubicin, Investigator propose a study of combining nivolumab with induction therapy with cyclophosphamide and doxorubicin for nonsquamous NSCLC with PD-L1 expression less than 10%.

DETAILED DESCRIPTION:
Nivolumab is now the standard of care for second-line treatment of advanced squamous or nonsquamous non-small cell lung cancer (NSCLC) regardless of the tumor's expression of programmed death-1 ligand (PD-1L). The 2015 Food and Drug Administration approval cited results from the Open-Label Randomized Phase III Trial of Nivolumab Versus Docetaxel in Previously Treated Metastatic nonsquamous-NSCLC (CheckMate057) trial. Those results showed that in unselected patients with advanced or recurrent nonsquamous NSCLC who had stopped responding to a platinum-based chemotherapy regimen, treatment with nivolumab produced significantly better overall survival during follow-up as long as 18 months, compared with a docetaxel-based regimen. But a more detailed assessment of the survival data showed an unexpected pattern of an early hazard among the nivolumab patients. During the first 3 months on randomized treatment, 15 more patients died in the nivolumab arm than in the docetaxel arm. This quickly reversed during months 4-6 on treatment, when nine more patients died on docetaxel than on nivolumab. By 12 months after the onset of treatment, overall survival was 51% in the nivolumab group and 39% among those randomized to docetaxel. A post hoc analysis showed a trend to a higher risk for death during the first 3 months of nivolumab treatment among patients with poorer prognostic features, more aggressive disease, and low or no tumor expression of PD-L1. In addition, only a subgroup of patients benefits from nivolumab with response rates of 20% in unselected cohorts and 10% in low PD-L1 expression cohort. Strategies to render the tumor micro-environment (TME) more susceptible to anti-PD1 might include stimulation of anti-cancer immune responses by induction treatment with low dose chemotherapy.

Cyclophosphamide, an old-school chemotherapeutic agent used across a wide range of malignancies, was found to be a potent immune modulator that targets suppressive regulatory immune cells within the tumor microenvironment while enhancing effector cells. However, cyclophosphamide has a limited effect on TIL from tumors larger than a few mm diameter in view of an increased percentage of myeloid derived suppressor cells (MDSC). Meanwhile, doxorubicin is also has a potent immune-modulating activity, which can selectively impair MDSC-induced immunosuppression. Additionally, both cyclophosphamide and doxorubicin have anti-tumor activity against NSCLC. Given the potent immune-modulating effects and anti-tumor activity of cyclophosphamide and doxorubicin, Investigator propose a study of combining nivolumab with induction therapy with cyclophosphamide and doxorubicin for nonsquamous NSCLC with PD-L1 expression less than 10%.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of nonsquamous NSCLC with SP263 PD-L1 expression <10%
* Patients whose tumor is not known to have anaplastic lymphoma kinase(ALK) or epidermal growth factor receptor(EGFR) mutation and Previously treated with at least one platinum-based chemotherapy but less than 3 prior chemotherapy
* Before study entry, a minimum of 21 days must have elapsed since any prior chemotherapy.
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
* No other forms of cancer therapy, such as immunotherapy for at least 2 weeks before the enrollment in study.
* Performance status of 0-1 on the ECOG criteria.
* At least one unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors (Revised RECIST guideline version 1.1)
* Estimated life expectancy of at least 8 weeks.
* Patient compliance that allow adequate follow-up. Adequate hematologic (WBC ≥4,000/mm3 또는 4.0 x 103/㎕ Platelet count ≥130,000mm3 또는 130 x 103/㎕ Bilirubin total ≤1.0 mg/dL AST/ALT≤ 80 IU/L creatinine concentration 1XULN or creatinine clearance (CrCl) > 50 mL/min (measured using the Cockcroft-Gault formula)
* Informed consent from patient or patient's relative.
* Males or females at least 18 years of age.

Exclusion Criteria:

* Previous therapy with anti-PD-1 or -PD-L1 inhibitors
* Persistence of clinically relevant therapy related toxicities from previous chemotherapy and/or radiotherapy
* Has received prior chemotherapy or tyrosine kinase inhibitor therapy within 3 weeks of the first dose of trial treatment ; completed palliative radiotherapy(except for brain and extremities) within 2weeks of the first dose of trial treatment. Prior curative thoracic radiation therapy(>=60Gy) is permitted if disease progression occured >4weeks after the completion of therapy.
* Treatment with other investigational drugs or treatment in another clinical trial within the past three weeks before start of therapy or concomitantly with this trial
* Has received a live vaccine(Concomitant yellow fever vaccin) within 4 weeks prior to the first administration of study medication. Concomitant yellow fever vaccination
* Active CNS metastases
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for 2 weeks prior to randomization
* Leptomeningeal disease
* Significant cardiovascular diseases (i.e., hypertension not controlled by medical therapy, unstable angina, history of myocardial infarction within the past 12 months, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion)
* Proteinuria CTCAE grade 2 or greater
* Significant weight loss (> 10 %) within the past 6 weeks prior to treatment in the present trial
* Current peripheral neuropathy ≥ CTCAE(version4.0) Grade 2 except due to trauma
* Major injuries and/or surgery with incomplete wound healing within the past ten days prior to enrollment
* Serious infections requiring systemic antibiotic (e.g. antiviral, antimicrobial, antifungal) therapy
* Active hepatitis C and/or B infection
* Known human immunodeficiency virus (HIV) seropositivity
* Serious illness or concomitant non-oncological disease such as neurologic-,psychiatric-, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least 7 months after end of active therapy
* Pregnancy or breast feeding
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
* Patients unable to comply with the protocol
* Active alcohol or drug abuse
* Other malignancy within the past three years other than basal cell skin cancer or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
objective response | From date of first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48months
  objective response rate using RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ji-youn han, Ph.D, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No